CLINICAL TRIAL: NCT06138288
Title: The Effect of Acupressure Applied After Cesarean Section on Postpartum Pain and Postpartum Comfort: A Randomized Controlled Study
Brief Title: Acupressure Applied After Cesarean Section on Postpartum Pain
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Hilal Begüm Çayır, Nurse, Eastern Mediterranean University
Other Study IDs: ETK00-2023-0107
Record Dates: First submitted 2023-07-19; First posted 2023-11-18 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Postpartum Disorder; Cesarean Section Complications
Keywords: cesarean section; acupressure; postpartum; pain; postpartum comfort
MeSH Terms: conditions — Puerperal Disorders; Pain | interventions — Acupressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- acupressure group: Women who are in acupressure will apply the application after cesarean section 2nd hour after applying the data collection forms (descriptive features formula, VAS, WHO). For women on acupressure, the application will be applied manually to the SP6, P6 and L14 points in the order indicated by the drawing with the index or middle finger, 1-1.5 cm depth for 5 seconds, pressing for 5 seconds, resting for 2 seconds and continuing for 2 minutes to go. will be with you. VAS will be filled again after the application.
  Interventions: Behavioral: acupressure
- control group

INTERVENTIONS:
Behavioral: acupressure — The acupressure points to be used in the research are located on the inner side of the lower leg, 4 fingers above the ankle and on the spleen meridian behind the tibia (SP6), which was previously effective in reducing pain, and located three fingers above the wrist (in the middle of the 2nd metacarpal bone, on the dorsum of the hand, adjacent The points determined as P6 (located between the metacarpal bones) and LI4 located in the space between the thumb and index finger (between the 1st and 2nd metacarpal bones of the hand, in the middle of the 2nd metacarpal bone on the radial side) were applied by a certified researcher to women in the acupressure group. will be done
  Groups: acupressure group

SUMMARY:
Pressure applied according to the principles of acupressure limits the pain limit, reduces the secretion of endorphins, which is a neurochemical, reduces the tension in the muscles, reduces the amount of oxygen in the blood flow, and finally provides duration and relaxation. Acupressure application is becoming more and more common nowadays because it is a noninvasive, safe, easy-to-apply and effective method without side effects. It seems that there is a limit to the study in which group acupressure applications in the literature are examined together on pain and comfort after cesarean section. In these basic points, the expectations of achieving postpartum pain and postpartum comfort of acupressure applied after cesarean delivery in this study. The circle of the research; There will be women who will have repeated cesarean section in a private Obstetrics Clinic in Famagusta. Women will be separated from two groups, one group will continue acupressure and the other group will do routine care. Visual analog scale and end-of-birth comfort procedure will be applied to women before and after the application.

DETAILED DESCRIPTION:
Pressure applied according to the principles of acupressure limits the pain limit, reduces the secretion of endorphins, which is a neurochemical, reduces the tension in the muscles, reduces the amount of oxygen in the blood flow, and finally provides duration and relaxation. Acupressure application is becoming more and more common nowadays because it is a noninvasive, safe, easy-to-apply and effective method without side effects. It seems that there is a limit to the study in which group acupressure applications in the literature are examined together on pain and comfort after cesarean section. In these basic points, the expectations of achieving postpartum pain and postpartum comfort of acupressure applied after cesarean delivery in this study. The circle of the research; There will be women who will have repeated cesarean section in a private Obstetrics Clinic in Famagusta. Women will be separated from two groups, one group will continue acupressure and the other group will do routine care. Visual analog scale and end-of-birth comfort procedure will be applied to women before and after the application.

ELIGIBILITY:
Inclusion Criteria:

* agreeing to participate in the research,
* be between the ages of 18-49,
* To give birth by cesarean section between 37-40 weeks,
* Having a healthy and live birth at the end of a single pregnancy,
* Receiving spinal anesthesia
* Being able to read and write Turkish and be open to communication.

Exclusion Criteria:

* Absence of pain in the 2nd hour postpartum
* Having a cesarean delivery after a risky pregnancy,
* Having a chronic illness
* Having severe systemic disease
* Not receiving spinal anesthesia
* Having a body mass index over 25,
* Have previous acupressure experience.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: 18-49 age women
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 5 minutes
  VAS has been developed to convert some values that cannot be measured numerically into numeric values. The VAS, which is a generally accepted, safe and easily applicable measurement tool in the world literature, consists of a 10 cm long line and there are subjective descriptive statements at both ends of the scale (0 cm = no pain and 10 cm = unbearable pain). The individual marks the appropriate place for his/her pain on this 10 cm line on the scale. The distance from the beginning of the scale to the point where the individual marks is measured with a ruler, and the pain intensity of the individual is determined numerically in cm. A low score obtained from the VAS indicates that the individual's pain intensity is low/low, and a high score indicates high/severe. The VAS is sensitive to pharmacological and non-pharmacological modalities that alter the pain experience.

SECONDARY OUTCOMES:
postpartum comfort scale | 15 minutes
  It was developed by Karakaplan and Yıldız (2010) to determine postpartum comfort. The scale is likert type and consists of 34 items. Each item is scored between "strongly agree" (5 points), and "strongly disagree" (1 point). I totally agree with positive sentences shows the best comfort (5 points), and negative sentences show low comfort (1 point). Accordingly, the lowest score to be taken from the scale is 34, and the highest score is 170. The scale has three sub-dimensions as "physical, psychospiritual and sociocultural". An increase in the score obtained from the scale indicates an increase in comfort. The Cronbach Alpha reliability of the scale was found to be .78 for the total DSQ.

CONTACTS AND LOCATIONS:
Locations (1):
- Hilal Begum Cayır, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cayir HB, Abic A. The effect of acupressure on postpartum pain and comfort after cesarean delivery: a randomized controlled trial. Women Health. 2024 Nov-Dec;64(10):892-903. doi: 10.1080/03630242.2024.2428793. Epub 2024 Nov 12. PMID 39532534